CLINICAL TRIAL: NCT05264259
Title: New Therapeutic Approach Against BK Virus Infection Based on Monoclonal Antibodies
Acronym: AcMBK
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8521
Record Dates: First submitted 2022-02-07; First posted 2022-03-03 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: BK Virus Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BK virus (BKV) infection has a major negative impact on transplant recipients. No BKV-specific antiviral therapy is available, so there is an urgent need to develop new anti-BKV preventive and therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* BK positive
* adult
* ok to participed to research

Exclusion Criteria:

* under guardianship
* under curatorship
* opposed to research
* deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adult patient with a posititive serology BK confirmed
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Ability of the isolated monoclonal antibodies to neutralize all 3 BKV genotypes | 5 years
  The neutralization titer will be defined as the dilution of the sample that produced 50% inhibition of pseudovirion infectivity (IC50)

CONTACTS AND LOCATIONS:
Overall Officials: Samira FAFI-KREMER, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service de Virologie - CHU Strasbourg - France, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided